CLINICAL TRIAL: NCT01150617
Title: Effect of Normalization of Fasting Glucose by Intensified Insulin Therapy on the Incidence of Restenosis After Peripheral Angioplasty in Patients With Type 2 Diabetes.
Brief Title: Normalization of Fasting Glucose and the Incidence of Restenosis After Peripheral Angioplasty
Acronym: LIMBISCH
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: end-point reached
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, PierMarco Piatti, PI, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Limb ischemia
Record Dates: First submitted 2010-06-23; First posted 2010-06-25 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Type 2 Diabetes Mellitus; Peripheral Vascular Disease
Keywords: Type 2 diabetes mellitus; Normoglycemia; Peripheral angioplasty
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Peripheral Vascular Diseases | interventions — Insulin Glargine; Hypoglycemic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- long-acting insulin plus analogues (Active Comparator): three administrations of regular insulin or short acting insulin analogues before meals combined with long-acting insulin analogue glargine in the evening.
  Interventions: Drug: Insulin glargine plus insulin analogues
- long-acting insulin and oral agents (Active Comparator): treatment will be once-daily long-acting insulin and oral antidiabetic agents
  Interventions: Drug: Insulin glargine plus insulin analogues

INTERVENTIONS:
Drug: Insulin glargine plus insulin analogues — * Intensified insulin therapy: three administrations of regular insulin or short acting insulin analogues before meals combined with long-acting insulin analogue glargine in the evening. The treatment goal will be a fasting blood glucose level of 5.5 mmol/L (99 mg/dl) and a HbA1c<6.5% at the end of the follow-up.
  * Standard care: treatment will be once-daily long-acting insulin and oral antidiabetic agents to achieve HbA1c levels of < 7.0% at the end of the follow-up.
  Other Names: Insulin glargine plus short acting insulin analogues; Insulin glargine plus hypoglycemic agents

SUMMARY:
Primary objective of the study is to test whether an intensified insulin therapy incorporating the target of normal fasting glucose (<5.5 mmol/L) and glycated hemoglobin <6.5% is able to halve the incidence of angiographic restenosis at 6 months (expected rate 45%, to be reduced at 15%) after peripheral angioplasty compared with standard care to achieve a glycated hemoglobin <7.0% in patients with type 2 diabetes and limb ischemia.

Secondary objectives include the identification of markers associated with, and predictive of, restenosis and the investigation of the underlying pathophysiological background, with specific focus on the role of nitric oxide (NO), mechanisms of endothelial activation/apoptosis, inflammation and matrix remodeling risk profiles, candidate gene polymorphisms and endothelial progenitor cells evaluation.

Methodology: This is a randomized, open-label, clinical trial comparing two regimens of insulin therapy having as an outcome measure the incidence of angiographic restenosis at 6 months after peripheral angioplasty. Seventy consecutive patients with type 2 diabetes and peripheral arterial disease undergoing peripheral angiography and subsequent angioplastic procedure will be studied. Patients will be treated by intensive insulin therapy, based on three pre-prandial administrations of regular insulin or short acting insulin analogues combined with the long-acting insulin analogue glargine or standard care based on once-daily insulin and oral antidiabetics agents. Patients randomized to the intensive insulin therapy arm will be educated and followed up with daily measurements of fasting glucose and weekly phone contacts with the target of fasting glucose <5.5 mmol/L (99 mg/dl) to obtain glycated hemoglobin <6.5%. The control arm will be followed to achieve a target of glycated hemoglobin <7.0%. Life style recommendations, including diet and physical activity program, will be the same for the two arms. All patients will undergo three visits with physical examination and blood sampling, at baseline and at 2, 4 and 6 months after angioplasty. Moreover, patients on normal fasting glucose arm will be monitored by phone on weekly basis in order to test their adherence to therapeutic target.

DETAILED DESCRIPTION:
The principal objectives of this project are:

Objectives Primary Objectives

To determine the role of fasting normoglycemia achieved with long term (6 months) intensified insulin therapy in:

* Reduction of angiographic restenosis (> or=50%) after peripheral angioplasty
* Increase in the rate of primary clinical success at follow-up defined as continued relief of ischemic rest pain, reduction in severity of claudication with persistent hemodynamic success and/or symptomatic improvement of at least one category according to Rutherford criteria, healing of ulceration, and freedom from unplanned surgical amputation or bypass surgery
* Definition of the beneficial effect of normoglycemia in insulin mediated nitric oxide (NO) modulation of neointima formation through its action on inflammation and/or matrix remodelling Secondary Objectives
* To determine whether fasting normoglycemia achieved with intensified insulin therapy is able to reduce or avoid planned or unplanned major amputation as limb loss above the metatarsal level and minor amputation, as transmetatarsal amputation or removal of more distal parts of the lower extremity and/or the performance of less extensive amputation than initially intended through 6 months
* To evaluate the reduction of Major Adverse Cardiovascular Event (MACE) defined as the occurrence of death, or repeat target vessel revascularization
* To find new risk profiles of systematically detectable indices able to define the patients at the highest risk to develop restenosis
* To correlate angiographic and clinical indices of restenosis with endothelial activation/apoptosis, inflammation and matrix remodelling risk profiles
* To define the association of candidate genes variants and the degree of restenosis
* To understand the impact of fasting normoglycemia achieved with intensified insulin therapy on endothelial progenitor cells isolation and gene expression involved in the process of vascular repair and in the inhibition of neointimal hyperplasia

This is a randomized, open-label, clinical trial comparing two regimens of insulin therapy (intensified insulin therapy vs standard care) to determine if fasting normoglycemia achieved with intensified insulin therapy is able to reduce the incidence of angiographic restenosis at 6 months after peripheral angioplasty.

Seventy consecutive patients with type 2 diabetes mellitus and peripheral arterial disease (PAD) defined at angiographic evaluation and/or clinical manifestations, will be admitted to our Institute to undergo PTA procedure. After the procedure, suitable patients will be screened to enter the study.

One week following hospital discharge after PTA procedure, patients will return to the Diabetology Outpatients Clinic to be randomly assigned to receive intensified insulin therapy or standard care. Prestudy treatments could be diet alone, oral antidiabetic agents, or once-daily insulin and oral antidiabetic agents.

Two groups will be evaluated

* Intensified insulin therapy: three administrations of regular insulin or short acting insulin analogues before meals combined with long-acting insulin analogue glargine in the evening. The treatment goal will be a fasting blood glucose level of 5.5 mmol/L (99 mg/dl) and a HbA1c<6.5% at the end of the follow-up.
* Standard care: treatment will be once-daily long-acting insulin and oral antidiabetic agents to achieve HbA1c levels of < 7.0% at the end of the follow-up.

Routine visits will be scheduled after 1, 2, 4 weeks and then at 2, 4 and 6 months.

All patients will be asked to monitor blood glucose levels each morning and document hypoglycemia and 1-day six point glucose profiles (before and 2 h after breakfast, lunch and dinner) before each clinic visit.

In the intensified insulin therapy arm, patients will be contacted by telephone every week to target fasting glucose levels at 5.5 mmol/L through a titrated regimen.

The following titration regimen will be followed, according with (48):

Mean of self-monitored FPG values Increase of long-acting insulin dosage (UI) >180 mg/dl (>10 mmol/l) 8 140-180 mg/dl (7.8-10 mmol/l) 6 120-140 mg/dl (6.7-7.8 mmol/l) 4 100-120 mg/dl (5.6-6.7 mmol/l) 2 72-100 mg/dl ( 4.0-5.6 mmol/l) no changes <72 mg/dl (<4.0 mmol/l) decrease 2 Ethics Approval The protocol is in accordance with the guidelines contained in the "Declaration of Helsinki 2" and with the current national legislation.

The protocol, the site's informed consent form and any other written information provided to the patients prior to any enrollment will be approved by the local Ethics Committee and the principal investigator will take responsibility to ensure that this procedure will be followed. If, during the study, it is necessary to amend the informed consent form, the investigator will be responsible for ensuring the local Ethics Committees reviews and approves these amended documents before to enter new subjects into the study.

Discomforts of patients included in the studies are in all cases mild and temporary. Risks involved in participating in all the studies are limited. Considering the potential benefits related to preventing restenosis after peripheral angioplasty in diabetic patients, we believe that these investigations are justified.

Utilization of drugs in this project will be subject to Institutional and National Safety Regulations to ensure the safety of workers and to prevent damage to the environment and community.

Experimental design During the hospitalization period, before procedure, from patients suitable to enter into the study, blood samples will be drawn before breakfast for evaluation of plasma glucose, serum insulin and plasma FFA. Samples will be drawn to evaluate gene polymorphisms, circulating endothelial progenitor cells isolation and to study insulin-mediated nitric oxide signalling pathway.

At the time of angiographic and angioplastic procedure, blood samples will be drawn from femoral arterial and venous districts for the evaluation of indices of endothelial activation/apoptosis, inflammation and matrix remodelling. A venous sample will be taken for endothelial progenitor cells isolation and gene expression evaluation.

After the procedure of peripheral angiography and angioplasty, in Outpatient Clinic, before randomisation, all patients will perform a baseline physical examination and blood samples to evaluate both the metabolic parameters to define the degree of glucose control and indices of endothelial activation/apoptosis, inflammation and matrix remodelling and DNA isolation.

At the time of this visit, patients will be randomly assigned to intensive insulin treatment for 6 months or to standard care for glycemic control, added to their usual cardiovascular treatment. A similar diet and physical activity program will be planned for both groups. At 2, 4 and 6 months, a physical examination and blood samples to evaluate both the metabolic parameters to define the degree of glucose control and indices of endothelial activation/apoptosis, inflammation and matrix remodelling will be repeated. Samples will be drawn to evaluate circulating endothelial progenitor cells and to study insulin-mediated nitric oxide signalling pathway and its modulation by prolonged strict fasting normoglycemia.

After 6 months or before in the presence of symptoms, they will perform an angiographic control and evaluated for the presence of restenosis. At this time, blood samples will be drawn from femoral arterial and venous districts for the evaluation of indices of endothelial activation/apoptosis, inflammation and matrix remodelling. A venous sample will be taken for endothelial progenitor cells isolation and gene expression evaluation. During the hospitalization period,blood samples will be drawn before breakfast for evaluation of plasma glucose, serum insulin and plasma FFA.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders
2. Age between 30 and 75 years
3. Early type 2 diabetes, defined as FPG >7.0 mmol/l or a PPG of 11.1 mmol/l or greater or a previous diagnosis of diabetes
4. Treatments accepted

   * Diet without pharmacological treatment
   * One or more oral antidiabetic drug (OAD: sulfonylureas, biguanides, meglitinides) at half-maximum dose or greater
   * Once daily insulin and OAD
5. Angiographic documentation of infrapopliteal arterial disease (stenosis >70% or occlusion)
6. Critical limb ischemia (CLI) defined as

   * Persistent, recurring rest pain requiring analgesia and an ankle systolic pressure <50 mm Hg and/or toe systolic pressure <30 mm Hg or TcPO2 <30 mm Hg
   * Ulceration, gangrene, or nonhealing wounds of the foot with ankle systolic pressure <50 mm Hg or toe systolic pressure <30 mm Hg or TcPO2 <30 mm Hg
   * Fontaine stages III-IV and rutherford categories IV-VI
   * Lifestyle-limiting claudication defined as Rutherford category II to III associated with jeopardized single vessel runoff or complete trifurcation vessel occlusion.
7. Subject able to provide a signed and dated written informed consent

Exclusion Criteria:

1. Type 1 diabetes, defined as positivity for GAD antibodies measured by radiobinding assay
2. Unwilling to inject insulin or to perform a correct self monitoring of blood glucose
3. Acute limb ischemia
4. Buerger disease
5. Severe contrast allergy
6. Hypersensitivity to aspirin and/or clopidogrel
7. Systemic coagulopathy contraindicating antiaggregation therapy
8. Hypercoagulation disorder
9. Serum creatinine>2.0 mg/dl at screening
10. Active liver disease, or ALT or AST >2.5 times upper limit of normal at screening
11. Chronic or recurrent treatment with systemic corticosteroids
12. Malignant diseases
13. Psychiatric diseases which make participation impossible
14. Alcohol abuse

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-12; Primary Completion 2010-11 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Reduction of restenosis after peripheral angioplasty | 6 months, average up to 30 weeks
  Primary objective of the study is to test whether an intensified insulin therapy incorporating the target of normal fasting glucose (<5.5 mmol/L) and glycated hemoglobin <6.5% is able to halve the incidence of angiographic restenosis at 6 months (expected rate 45%, to be reduced at 15%) after peripheral angioplasty compared with standard care to achieve a glycated hemoglobin <7.0% in patients with type 2 diabetes and limb ischemia.

SECONDARY OUTCOMES:
Identification of new peripheral markers predictive of restenosis | 6 months, average up to 30 weeks
  Secondary objectives include the identification of markers associated with, and predictive of, restenosis and the investigation of the underlying pathophysiological background, with specific focus on the role of nitric oxide (NO), mechanisms of endothelial activation/apoptosis, inflammation and matrix remodeling risk profiles, candidate gene polymorphisms and endothelial progenitor cells evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: PierMarco Piatti, MD, Principal Investigator — San Raffaele Scientific Institute, Milan
Locations (1):
- Cardio-Metabolic and Clinical Trials Unit, San Raffaele Scientific Institute, Milan, Italy